CLINICAL TRIAL: NCT01574261
Title: Could the Therapy With Inositol Affect the Cardiovascular Risk in PCOS Women? Results of a Randomized Clinical Trial
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Rosanna Apa, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: disfunzionale12
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Cardiovascular risk; Metabolic Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Metabolic Syndrome | interventions — Inositol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inositol (Active Comparator): Patients will be randomized to receive Inositol 4 g/die per os for four months of treatment
  Interventions: Drug: Inositol
- Placebo (Placebo Comparator): Patients will be randomized to receive placebo for four months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo for four months
  Arms: Placebo
Drug: Inositol — Inositol 4g/die for four months
  Arms: Inositol

SUMMARY:
Polycystic ovary syndrome (PCOS) is associated with an increased cardiovascular risk. The aim of the study was to evaluate long-term effects of inositol on some cardiovascular risk factors in PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic Ovary Syndrome
* Age >18 and <35

Exclusion Criteria:

* Chronic or acute inflammatory disease, cancer, autoimmune disease, treatment during the last 6 months prior to our evaluation, DM2, hypertension, major surgery in the last 3 months or other hormonal dysfunctions (hypothalamic, pituitary, thyroidal, or adrenal causes).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
CD4+ CD28 null T-lymphocyte frequency | five minutes

SECONDARY OUTCOMES:
insulinaemic area OGTT AUCi, lipid profile, androgen levels | 120 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Università cattolica S. Cuore, Rome, Rome, Italy

REFERENCES:
- [Result] Niccoli G, Apa R, Lanzone A, Liuzzo G, Spaziani C, Sagnella F, Cosentino N, Moro F, Martinez D, Morciano A, Baca M, Pazzano V, Gangale MF, Tropea A, Crea F. CD4+CD28 null T lymphocytes are expanded in young women with polycystic ovary syndrome. Fertil Steril. 2011 Jun 30;95(8):2651-4. doi: 10.1016/j.fertnstert.2011.01.129. Epub 2011 Feb 16. PMID 21324454